CLINICAL TRIAL: NCT04518254
Title: Contribution of L-Tyrosine to Human Decision Making in Stressful Situations
Acronym: TYRO-STRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018PPRC25; 2019-A03194-53 (Other: IDRCB)
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Stress, Psychological
Keywords: L-tyrosine
MeSH Terms: conditions — Stress, Psychological | interventions — Blood Specimen Collection; Tyrosine; Electromyography; Electroencephalography

STUDY DESIGN:
Intervention Model Description: The study is composed of 4 arms:
  1. Tyrosine treatment without stress exposure
  2. Tyrosine treatment with stress exposure
  3. Placebo treatment without stress exposure
  4. Placebo treatment with stress exposure
  Every participants will participate in the 4 arms in a random order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The pharmacist, carrying out the packaging and labelling of the treatment units, will ensure the blinding. Neither the participant nor the investigator will know what treatment is being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tyrosine - Test (Experimental): 4 similar visits (day 0, day 3, day 6, day 9): Administration of L-tyrosine No stress exposure
  Interventions: Biological: Blood collection; Drug: L-Tyrosine 500 Mg; Behavioral: Cognitive tasks; Behavioral: Anxiety scale; Device: Electromyography (EMG); Device: Electroencephalography (EEG)
- Tyrosine - Stress (Experimental): 4 similar visits (day 0, day 3, day 6, day 9): Administration of L-tyrosine Stress exposure
  Interventions: Biological: Blood collection; Drug: L-Tyrosine 500 Mg; Behavioral: Cognitive tasks; Other: Stress exposure; Behavioral: Anxiety scale; Device: Electromyography (EMG); Device: Electroencephalography (EEG)
- Placebo - Test (Experimental): 4 similar visits (day 0, day 3, day 6, day 9): Administration of Placebo No stress exposure
  Interventions: Biological: Blood collection; Drug: Placebo; Behavioral: Cognitive tasks; Behavioral: Anxiety scale; Device: Electromyography (EMG); Device: Electroencephalography (EEG)
- Placebo - Stress (Experimental): 4 similar visits (day 0, day 3, day 6, day 9): Administration of Placebo Stress exposure
  Interventions: Biological: Blood collection; Drug: Placebo; Behavioral: Cognitive tasks; Other: Stress exposure; Behavioral: Anxiety scale; Device: Electromyography (EMG); Device: Electroencephalography (EEG)

INTERVENTIONS:
Biological: Blood collection — A blood sample will be collected before and after treatment administration
Drug: L-Tyrosine 500 Mg — The participants will be administered 4 capsules of L-Tyrosine 500 mg per oral route
  Arms: Tyrosine - Stress; Tyrosine - Test
Drug: Placebo — The participants will be administered 4 capsules of Lactose 500 mg (placebo) per oral route
  Arms: Placebo - Stress; Placebo - Test
Behavioral: Cognitive tasks — The participants will perform cognitive decision-making tasks: Simon task and masking task after treatment administration
Other: Stress exposure — Unpleasant but not painful skin stimulations will be administered to the participants at variable intervals on the left leg during the cognitive tasks
  Arms: Placebo - Stress; Tyrosine - Stress
Behavioral: Anxiety scale — Spielberger's State Trait Anxiety Inventory (STAI) will be filled by the participants before and after cognitive tasks
Device: Electromyography (EMG) — Electromyography measurements will be performed during cognitive tasks.
Device: Electroencephalography (EEG) — Electroencephalography measurements will be performed during cognitive tasks.

SUMMARY:
L-tyrosine is a chemical precursor of dopamine. Under specific conditions, tyrosine administration can increase brain dopamine levels and therefore several studies have explored whether tyrosine supplementation can have a beneficial effect on cognitive and behavioural performance that is dependent on dopaminergic function. However, the effects of tyrosine supplementation are mixed: some studies show positive effects while others do not. Stress leads to an increase in dopaminergic activity and turnover in the brain, resulting in a decrease in brain dopamine levels. We propose to study the contribution of tyrosine to decision making and more particularly to the processes of response selection (mediated by the prefrontal cortex and under the influence of the dopaminergic system) in stressful situations.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 65 years of age

Exclusion Criteria:

* Tyrosine intake within the previous 15 days
* History of neurological or psychiatric disorder
* History of nephrological or endocrine disorder or liver failure
* Hereditary tyrosinemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Reaction Time | At day 9 (9 days after enrollment)
  Reaction Time at the cognitive tasks
Number of incorrect responses | At day 9
  Number of incorrect responses at the cognitive tasks

SECONDARY OUTCOMES:
Error negativity | At day 9
  Error negativity on motor evoked potentials (measured by EMG)
Correlation coefficient between anxiety level and tyrosinemia | At day 9
  Correlation coefficient between anxiety level (measured by anxiety scale) and tyrosinemia (measured in blood sample)
Correlation coefficient between anxiety level and plasma tyrosine | At day 9
  Correlation coefficient between anxiety level (measured by anxiety scale) and plasma tyrosine (measured in blood sample)
Correlation coefficient between cortisolaemia and melatoninaemia | At day 9
  Correlation coefficient between cortisolaemia and melatoninaemia (measured in blood sample)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided